CLINICAL TRIAL: NCT01354704
Title: Echo-Doppler Assessment of the Occurrence of Asymptomatic Deep Vein Thrombosis (DVT) in Orthopedic Replacement Surgery Under Enoxaparine (PRENOXA)
Brief Title: Echo-Doppler Assessment of the Occurrence of Asymptomatic DVT in Orthopedic Replacement Surgery Under Enoxaparin
Acronym: PRENOXA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Les Laboratoires des Médicaments Stériles (Industry)
Collaborators: Hopital Charles Nicolle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PRENOXA_2011
Record Dates: First submitted 2011-05-14; First posted 2011-05-17 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2012-02

CONDITIONS: Deep Vein Thrombosis; Venous Thrombosis; Adverse Effect of Anticoagulants
Keywords: deep veinous thrombosis; enoxaparin
MeSH Terms: conditions — Venous Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- lovenox (Active Comparator): patient under lovenox 4000 IU
  Interventions: Drug: Enoxaparin
- enoxa (Active Comparator): patients under Enoxa 4000 IU
  Interventions: Drug: Enoxaparin
- total knee replacement (No Intervention): patients undergoing total knee replacement
- total hip replacement (No Intervention): patient undergoing total knee replacement

INTERVENTIONS:
Drug: Enoxaparin — enoxaparin 4000 IU 1 injection/day in subcutaneous.
  Arms: enoxa; lovenox

SUMMARY:
The objectives of the study are:

o Objective ultrasound: Determine the presence or absence of subclinical DVT in practicing ultrasound-Doppler Day7 and Day35, patients who underwent TKA or THA

o Clinical objective To evaluate the efficacy and tolerability clinical Enox ® in these patients compared with the original drug Lovenox ®.

ELIGIBILITY:
Inclusion Criteria:

* man or woman aged over 18 years, admitted to undergo orthopedic total knee or total hip prosthesis requiring the use of enoxaparin 4000 IU for the Prophylaxis.

Exclusion Criteria:

* Patient participating in another study.
* hypersensitivity to enoxaparin sodium, heparin unfractionated heparin or other low molecular weight.
* Patients at risk of major bleeding or uncontrolled including patients with recent stroke
* Pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2011-03; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Presence or absence of ultrasound findings in favor of asymptomatic DVT | Day 7 and 35
  After orthopedic surgery, patients are put under LMWH thromboprophylaxis based but some patients may be carrying an asymptomatic DVT. so we'll try the distal venous thrombosis rate in these patients using Doppler ultrasound.

SECONDARY OUTCOMES:
To evaluate the efficacy and tolerability clinical Enox ® in these patients. | 3 months
  Criteria for evaluating the effectiveness of Enox ®:
  * Onset or without clinical signs of deep vein thrombosis in clinical postoperative
  * Onset or without clinical signs of pulmonary embolism after surgery

CONTACTS AND LOCATIONS:
Overall Officials: mondher kooli, MD, Study Chair — Hospital Charles Nicolle; Ramzi Bouzidi, MD, Principal Investigator — Hospital Charle Nicolle; Mustapha Azaiz, MD, Principal Investigator — Delta Medical Center; Abdelaziz Zarrouk, MD, Principal Investigator — Hospital Charles Nicollle
Locations (1):
- Hospital Charle Nicolle, Tunis, Tunis BAB Souika, Tunisia

REFERENCES:
- [Result] 1- Physiopathologie et prévention de la maladie thromboembolique veineuse postopératoire. Charles Marc Samama, Pierre Albaladejo. Sang Thrombose Vaisseaux 2008 ; 20, n°3 :138-43 2- Thromboses veineuses profondes. Dr Jean - Marc Schleich. Département de cardiologie et maladies vasculaires ; CHU de Rennes ; mis à jour le 6 septembre 1998 3- Prévention de la Thrombose veineuse. Dr H. Raybaud - MAJ 2006. Esculape.com : site de médecine générale. 4- Thrombose veineuse profonde. J. - L. Bosson, A. Franco. 1995 SIIM CHU de Grenoble 5- Suivi écho-doppler de thromboses veineuses profondes distales asymptomatique. M.-T BARRELLIER et col. Journal des maladies vasculaires. Masson, 2000, 25, 3 195-200. 6- 83ème Réunion annuelle de la société française de chirurgie orthopédique et traumatologique. Résumé des communications. Revue de chirurgie orthopédique et réparatrice de l'appareil moteur (2008) 94S, S231-S327.